CLINICAL TRIAL: NCT03046628
Title: A Feasibility Study of Using Technology Based on Polarized Laser Light and Speed Camera for Non-invasive Tissue Perfusion Assessment of the Lower Extremities
Brief Title: Evaluation of Lower Extremity Tissue Perfusion With Polarized Laser Light
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC1602-16CTIL
Record Dates: First submitted 2017-01-10; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Ulcer; Perfusion

ARMS (1):
- Patients with diabetic feet ulcers (Experimental): Each patient will be examined twice, first with TcPO2 (TCM400, Radiometer Medical ApS, Denmark) and then with a green laser (harmonic of continuous neodymium-doped yttrium aluminium garnet laser 532-nm wavelength and fast camera (PixelLink PLE531) system.
  Interventions: Device: TcPO2; Device: Green laser (at 532nm) and a fast camera

INTERVENTIONS:
Device: TcPO2
  Other Names: TCM400, Radiometer, Denmark
Device: Green laser (at 532nm) and a fast camera
  Other Names: PixelLink PL-E531, continuous green laser

SUMMARY:
The aim of this study is to test the feasibility of using polarised green laser and CMOS camera in order to assess the tissue perfusion of lower extremity ulcers in patients suffering from diabetic foot by comparing this method with the percutaneous tissue oxygen tension examination which is currently the "gold standard" examination.

DETAILED DESCRIPTION:
An objective assessment of blood supply and oxygen delivery to the damaged tissue in patients with diabetic ulcer is very problematic with various currently accepted auxiliary examinations. These tests include measuring blood pressure ratio between the ankle or toes arm (ABI \ TBI), Sonar Doppler examination of the lower limb arteries, and percutaneous tissue oxygen tension examination (TcPO2). Each of these tests, along with the obvious advantages esprit ability to assess a non-invasive blood as number of disadvantages.

As the blood supply to the tissue is the most important healing of the tissue regardless of the type of intervention chosen (conservative treatment includes systemic antibiotics or surgical debridement), there is clear necessity for a non-invasive test with high reliably assessing tissue perfusion in patients with diabetic ulcers.

Recently, a new a method for assessing multiple features in vital tissues using polarised laser light was introduced. The technique is based on tracking temporal changes of reflected secondary speckles produced in the skin when being illuminated by a laser beam. Change in skin's temporal vibration profile is generated by time varied oxygen concentration caused these temporal changes. This technology of nanometer motion sensing allows, according to studies already carried out, monitoring parameters such as blood pressure, pulse rate and heart rhythm, glucose concentration in the blood substances and alcohol, oxygen saturation and intraocular pressure.

In this study the investigators will examine, non-invasively, the tissue around the lower limb ulcers of 30 diabetic patients, beginning with the TcPO2 examination followed by the polarised laser light and complementary metal-oxide semiconductor (CMOS) camera examination, and analysing the data in order to determine the ability of the latter method for assessing the tissue oxygen pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic diabetic ulcers

Exclusion Criteria:

* Patients after amputation of some part in the lower limb
* Patients with acute infection on bony involvement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between TcPO2 results and reflected secondary speckle patterns | through study completion, an average of 1 year
  recording and comparing between the examinations of each diabetic ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Meir Nyska, Prof., Study Director — Head of the orthopaedic department

REFERENCES:
- [Background] LoGerfo FW, Coffman JD. Current concepts. Vascular and microvascular disease of the foot in diabetes. Implications for foot care. N Engl J Med. 1984 Dec 20;311(25):1615-9. doi: 10.1056/NEJM198412203112506. No abstract available. PMID 6390204
- [Background] Consensus development conference on diabetic foot wound care. 7-8 April 1999, Boston, MA. American Diabetes Association. Adv Wound Care. 1999 Sep;12(7):353-61. No abstract available. PMID 10687555
- [Background] Rayman G, Williams SA, Spencer PD, Smaje LH, Wise PH, Tooke JE. Impaired microvascular hyperaemic response to minor skin trauma in type I diabetes. Br Med J (Clin Res Ed). 1986 May 17;292(6531):1295-8. doi: 10.1136/bmj.292.6531.1295. PMID 2939920
- [Background] Schaper NC, Andros G, Apelqvist J, Bakker K, Lammer J, Lepantalo M, Mills JL, Reekers J, Shearman CP, Zierler RE, Hinchliffe RJ. Diagnosis and treatment of peripheral arterial disease in diabetic patients with a foot ulcer. A progress report of the International Working Group on the Diabetic Foot. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:218-24. doi: 10.1002/dmrr.2255. PMID 22271741
- [Background] Alexandrescu VA, Hubermont G, Philips Y, Guillaumie B, Ngongang C, Vandenbossche P, Azdad K, Ledent G, Horion J. Selective primary angioplasty following an angiosome model of reperfusion in the treatment of Wagner 1-4 diabetic foot lesions: practice in a multidisciplinary diabetic limb service. J Endovasc Ther. 2008 Oct;15(5):580-93. doi: 10.1583/08-2460.1. PMID 18840046
- [Background] Lukkari-Rautiarinen E, Lepantalo M, Pietila J. Reproducibility of skin blood flow, perfusion pressure and oxygen tension measurements in advanced lower limb ischaemia. Eur J Vasc Surg. 1989 Aug;3(4):345-50. doi: 10.1016/s0950-821x(89)80072-6. PMID 2670609
- [Background] Beiderman Y, Amsel AD, Tzadka Y, Fixler D, Mico V, Garcia J, Teicher M, Zalevsky Z. A microscope configuration for nanometer 3-D movement monitoring accuracy. Micron. 2011 Jun;42(4):366-75. doi: 10.1016/j.micron.2010.05.020. Epub 2010 Sep 19. PMID 20888247
- [Background] Zalevsky Z, Beiderman Y, Margalit I, Gingold S, Teicher M, Mico V, Garcia J. Simultaneous remote extraction of multiple speech sources and heart beats from secondary speckles pattern. Opt Express. 2009 Nov 23;17(24):21566-80. doi: 10.1364/OE.17.021566. PMID 19997398
- [Background] Beiderman Y, Horovitz I, Burshtein N, Teicher M, Garcia J, Mico V, Zalevsky Z. Remote estimation of blood pulse pressure via temporal tracking of reflected secondary speckles pattern. J Biomed Opt. 2010 Nov-Dec;15(6):061707. doi: 10.1117/1.3505008. PMID 21198155
- [Background] Beiderman Y, Blumenberg R, Rabani N, Teicher M, Garcia J, Mico V, Zalevsky Z. Demonstration of remote optical measurement configuration that correlates to glucose concentration in blood. Biomed Opt Express. 2011 Mar 14;2(4):858-70. doi: 10.1364/BOE.2.000858. PMID 21483609
- [Background] Ozana N, Arbel N, Beiderman Y, Mico V, Sanz M, Garcia J, Anand A, Javidi B, Epstein Y, Zalevsky Z. Improved noncontact optical sensor for detection of glucose concentration and indication of dehydration level. Biomed Opt Express. 2014 May 22;5(6):1926-40. doi: 10.1364/BOE.5.001926. eCollection 2014 Jun 1. PMID 24940550
- [Background] Margalit I, Beiderman Y, Skaat A, Rosenfeld E, Belkin M, Tornow RP, Mico V, Garcia J, Zalevsky Z. New method for remote and repeatable monitoring of intraocular pressure variations. J Biomed Opt. 2014 Feb;19(2):027002. doi: 10.1117/1.JBO.19.2.027002. PMID 24503638
- [Background] Golberg M, Fixler D, Shainberg A, Zlochiver S, Mico V, Garcia J, Beiderman Y, Zalevsky Z. Speckle-based configuration for simultaneous in vitro inspection of mechanical contractions of cardiac myocyte cells. J Biomed Opt. 2013 Oct;18(10):101310. doi: 10.1117/1.JBO.18.10.101310. PMID 23856787